CLINICAL TRIAL: NCT05053100
Title: Hemorrhage and Thrombosis in Hematology Malignancies: Understanding the Risks of Thrombosis and Anticoagulation in Patients With Hematologic Malignancies (HAT Trial)
Brief Title: Understanding the Risk of Blood Clots and Bleeding in Patients With Hematological Malignancies, HAT Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC210804; NCI-2021-09154 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-006940 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Acute Leukemia; Deep Vein Thrombosis; Hematopoietic and Lymphoid Cell Neoplasm; Hodgkin Lymphoma; Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma; Plasma Cell Myeloma; Thrombocytopenia
MeSH Terms: conditions — Venous Thrombosis; Hematologic Neoplasms; Hodgkin Disease; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin; Multiple Myeloma; Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (record review, blood collection): Patients' electronic health record are reviewed for 12 months and/or undergo collection of blood at pretreatment and on days 7, 28, 90, and 180.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection
Other: Electronic Health Record Review — Undergo electronic health record review

SUMMARY:
This study evaluates the risks and experience of blood clots and bleeding in patients with blood cancers. While it is standard of care to use medications to reduce the risk of blood clots in hospitalized individuals, some patients with blood cancers have low platelet counts that can increase the concern for bleeding complications associated with these medications. At this time, the optimal management strategies for blood clots are not well known for patients with blood cancers. This pilot study evaluates additional information that could help doctors know which patients are at highest risk for blood clots.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the incidence of hemorrhage in the 3 months following deep vein thrombosis diagnosis in hospitalized malignant hematology patients, based on anticoagulant use and presence of thrombocytopenia.

II. Determine recurrent or progressive venous thromboembolism in the 3 months following deep vein thrombosis diagnosis in hospitalized malignant hematology patients, based on anticoagulant use and presence of thrombocytopenia.

SECONDARY OBJECTIVES:

I. Assess feasibility of database creation of patient and clinical characteristics regarding thrombosis and hemorrhage in hospitalized malignant hematology patients.

II. Assess feasibility of patient enrollment and hemostatic laboratory collection pre, during and post treatment.

III. Describe the impact of thrombocytopenia on resource utilization following thrombosis diagnosis (blood product administration, imaging studies performed, number of days hospitalized).

IV. Describe the impact of therapeutic anticoagulation vs prophylactic anticoagulation on resource utilization following thrombosis diagnosis (blood product administration, imaging studies performed, number of days hospitalized).

V. Define baseline hemostatic characteristics in hospitalized malignant hematology patients prior to chemotherapy and the association with thrombosis or hemorrhage.

VI. Describe changes in laboratory hemostatic characteristics pre-treatment, during treatment and post treatment.

OUTLINE:

Patients' electronic health record are reviewed for 12 months and/or undergo collection of blood at pretreatment and on days 7, 28, 90, and 180.

ELIGIBILITY:
Inclusion Criteria:

* All unique patients, age > 18 years old, admitted to the Mayo Clinic Arizona Hematology A and B Service for initiation of 1.) new (or next line) chemotherapy, 2.) autologous stem cell transplant, or 3.) allogeneic stem cell transplant for a hematologic malignancy

Exclusion Criteria:

* Solid tumor malignancy patients
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Mayo Clinic Arizona Hematology.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Thrombosis incidence | Up to 1 year
  Assessed by incidence of hemorrhage following deep vein thrombosis diagnosis, based on anticoagulant use and presence of thrombocytopenia
Rate of venous thromboembolism (VTE) recurrence | Up to 1 year
  Assessed as the time from admission to the hospital and Venous thrombotic event

SECONDARY OUTCOMES:
Hemorrhage incidence, without prior thrombosis | Up to 1 year
  Assessed as the time from admission to the hospital until hemorrhage incidence (without prior thrombosis)
Hemorrhage incidence, with prior thrombosis < 12 months | Within 3 months following deep vein thrombosis diagnosis
  Assessed as the time from admission to the hospital until Hemorrhage incidence (with prior thrombosis) < 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Leslie J. Padrnos, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials